CLINICAL TRIAL: NCT01014611
Title: Evaluation of Calcium Homeostasis and Mitochondrial Function in Skeletal Muscle in Subjects With Heart Failure, Before and After Exercise Training
Brief Title: Impact of Heart Failure on Calcium Homeostasis and Mitochondrial Function in Human Skeletal Muscle
Acronym: Calcicard
Status: Terminated | Type: Observational
Why Stopped: Difficulties of recruitement
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Ministry of Health, France (Other Government); National Cancer Institute, France (Other Government); Institut de Recherches Internationales Servier (Other)
Responsible Party: Sponsor
Other Study IDs: C08-23; 2008-A00936-49 (Registry Identifier: IDRCB)
Record Dates: First submitted 2009-11-16; First posted 2009-11-17 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-09

CONDITIONS: Heart Failure
Keywords: Heart failure; Skeletal muscle; Calcium; Ryanodine receptor; Mitochondria; Exercise training; Muscle biopsy; Healthy volunteers
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Class II NYHA Heart Failure: Fraction of ejection between 40% and 30%
- Class III NYHA Heart Failure: Fraction of ejection lower than 30%
- Healthy volunteers: Matched with patients on age and physical activity

SUMMARY:
The aim of this project is to investigate the impact of heart failure (HF) on calcium homeostasis, mitochondrial function and oxidative stress in human skeletal muscle, before and after exercise training. The role playing by circulating factors such as cytokines and catecholamines will also be evaluated.

24 HF patients will be enrolled in the study: 12 class II NYHA HF volunteers with a fraction of ejection between 40% and 30 %, and 12 class III NYHA HF volunteers with a fraction of ejection lower than 30 %. They will be compared to 24 sedentary healthy volunteers, matched on age and physical activity.

DETAILED DESCRIPTION:
Heart failure (HF) is associated with a skeletal muscle dysfunction, characterized by an increased fatigue that does not correlate with impaired myocardial function and physical inactivity that is commonly associated with HF. We identified in skeletal muscle of HF rats, a dysfunction of type 1 ryanodine receptors (RyR1) similar to that observed on the cardiac channel (RyR2), due to an hyperphosphorylation of the RyR and a dissociation of the regulatory protein FKBP12. This dysfunction, in addition to mitochondrial impairment, contributes in this animal model to the reduced exercise capacity observed during HF. Our goal is to analyse the impact of HF on calcium homeostasis, mitochondrial function and oxidative stress in human skeletal muscle. This project, performed on muscle biopsies, will also allow us to correlate calcium homeostasis and mitochondrial function (before and after exercise training) to circulating factors (cytokines, catecholamines) susceptible to trigger this muscle dysfunction.

This project addresses two straightforward questions about physiopathological mechanisms involved in skeletal muscle dysfunction during HF. To this aim we have built locally a network of laboratories and clinical services, used to work together, composed of two services of the University Hospital of Montpellier (Dept. of Cardiology and Dept of Clinical Physiology), an Inserm unit (U637, team 2) all interfaced by an another Inserm facility: the Clinical Investigation Center (CIC) of Montpellier. In this project we will focus on the dilated post-ischemic cardiomyopathy and compare two groups of patients under similar treatments studied at different stages of HF defined by the NYHA. The first patients (class II of NYHA) with a fraction of ejection between 40% and 30 % will be compared with patients (class III) with an ejection fraction lower than 30% (12 males, 35-65 years old per HF). 24 voluntary healthy sedentary individuals carefully selected for similar level of activity as for patients will be matched to the HF groups. All individuals will undergo cardiovascular explorations (ECG and echocardiography, blood test) at the inclusion. They will perform an exercise testing to evaluate their exercise capacity. A muscle biopsy will be performed 4 days after the exercise testing to assess the mitochondrial function and the Ca2+ homeostasis. After a rest period of 5 days, HF patients will perform a resistance-training program (3 times per week for 10 weeks). A 2nd cardiovascular explorations, exercise testing and muscle biopsy will then be performed to evaluate the beneficial effect of training. Mitochondrial function will be measured by oxygraphy and ATP production. Ca2+ homeostasis will be evaluated by confocal microscopy by recording spontaneous Ca2+ release events (i.e. RyR activity). Mitochondrial and RyR biochemical analysis will complete these functional studies as well as circulating factors (cytokines, catecholamine) and their associated receptors.

This project will allow us to characterize the behaviour of RyR in relation with mitochondrial function in human skeletal muscle during HF and identify beneficial effects of exercise training routinely proposed to HF patients. The analysis of circulating factors will allow us to establish a relation of cause and effect between myocardial dysfunction and muscle dysfunction. This project could thus open important perspectives in therapeutic. Compounds analogues to JTV-519, acting in stabilizing RyR channels, could be prescribed as a potent medication for HF. This project could thus be determinant in the comprehension of the regulation of Ca2+ and energetic metabolism in human skeletal muscle which could be an appropriate model to evaluate the effects of new pharmacological agents.

ELIGIBILITY:
Inclusion Criteria:

* BMI < 30

Exclusion Criteria:

* Contra-indication to exercise testing performance and muscle biopsy

Ages: 35 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 24 heart failure patients: 12 class II NYHA with a fraction of ejection between 40% and 30% and 12 class III NYHA with a fraction of ejection lower than 30% 24 sedentary healthy male volunteers matched to patients on age and physical activity
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2010-04; Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the skeletal muscular function (calcium homeostasis, mitochondrial function and oxidative stress) in two stages of heart failure patients compared to healthy volunteers | Baseline measurement

SECONDARY OUTCOMES:
To analyse the link between the hypothetical skeletal muscular function in two stages of heart failure and circulating factors such as cytokines and catecholamines | Baseline measurement
To investigate the effect of exercise training on skeletal muscular hypothetical dysfunction in two stages of heart failure patients | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Florence Galtier, MD, Principal Investigator — CHRU de Montpellier, France; Alain Lacampagne, PHD, Study Director — INSERM, France
Locations (1):
- Centre Hospitalier Régional Universitaire, Montpellier, France